CLINICAL TRIAL: NCT02852174
Title: Mindfulness-Based Stress Reduction for Wounded Warrior Caregivers
Brief Title: The Veteran Caregiver Reducing Stress Time (VetCareReST) Study
Acronym: VetCareReST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandraluz Lara-Cinisomo (Other)
Responsible Party: Sponsor-Investigator, Sandraluz Lara-Cinisomo, Assistant Professor, University of Illinois at Urbana-Champaign
Organization: University of Illinois at Urbana-Champaign (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16648
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Stress, Depression, Anxiety and Worry
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness group (Experimental): The treatment groups will participate in a mindfulness intervention training that will meet for 2 hours once a week for eight weeks. The 8-week program provides participants with 2-hour weekly instruction designed to teach specific skills and how to apply them during stressful situations (e.g., when caring for or advocating for the veteran).Mindfulness training also requires that participants engage in daily home practice for 30 to 40 minutes. Participants will be required to record the duration of the meditation in log sheets.
  Interventions: Behavioral: Mindfulness meditation training
- Control (No Intervention): Participants in the control may receive the mindfulness training after the wait period ends at which point they may receive the treatment as described above.

INTERVENTIONS:
Behavioral: Mindfulness meditation training — Mindfulness meditation training
  Arms: Mindfulness group

SUMMARY:
Caring for a disabled adult, particularly those with long-lasting impairment, has been associated with elevated levels of stress, depression and anxiety among caregivers.Recent studies show that veteran caregivers experience higher levels of psychological distress than caregivers in the general population, highlighting the psychological needs of this population. The Veteran Caregiver Reducing Stress Time (VetCareReST) is a randomized control trial designed to test the effectiveness of a mindfulness at reducing stress, depression and anxiety in veteran caregivers in Champaign and Danville County.

DETAILED DESCRIPTION:
Recent estimates indicate that there are 275,000 to one million informal veteran caregivers. Caring for a disabled adult, particularly those with long-lasting impairment, has been associated with elevated levels of stress, depression and anxiety among caregivers. Veteran caregivers are especially vulnerable because of competing demands. For instance, Post 9/11 veteran caregivers are more likely to be the spouse of a veteran, and have experienced the stress of multiple deployments, have a young child in their care, and work outside the home. Recent studies show that veteran caregivers experience higher levels of psychological distress than caregivers in the general population, highlighting the psychological needs of this population. One effective approach at reducing stress, depression and anxiety has been the use of mindfulness training, which has been shown to effectively reduce mood symptoms among professional caregivers. The Veteran Caregiver Reducing Stress Time (VetCareReST) is a randomized control trial designed to test the effectiveness of a mindfulness at reducing stress, depression and anxiety in veteran caregivers in Champaign and Danville County. This study builds on Dr. Lara-Cinisomo's (PI) experience with military spouses. The findings from this trial will serve as pilot data for a large-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Provide unpaid caregiver or support to a veteran
* Must be 18 years of age or older
* Willing to participate for the duration of the project
* Able to track his/her home practice in a handwritten log
* Have no significant psychiatric disorders other than depression or anxiety (e.g., bipolar disorder, substance abuse, actively suicidal)

Exclusion Criteria:

* The presence of significant psychiatric disorders other than depression or anxiety (e.g., bipolar disorder, substance abuse, actively suicidal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Stress | 8 weeks
  Perceived levels of stress

SECONDARY OUTCOMES:
Depressed mood | 8 weeks
  Depressive symptoms

OTHER OUTCOMES:
Anxiety | 8 weeks
  Anxious symptoms
Worry | 8 weeks
  Worried feelings

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States